CLINICAL TRIAL: NCT06032325
Title: Neutrophil Gelatinase Associated Lipocalin and Kidney Injury Molecule-1 As Biomarkers of Acute Kidney Injury in Children With Diabetic Ketoacidosis
Brief Title: Neutrophil Gelatinase Associated Lipocalin and Kidney Injury Molecule-1 As Biomarkers of AKI in Children With DKA
Acronym: AKI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bassem Eldaba Hosny Fares, resident, Assiut University
Other Study IDs: 1010
Record Dates: First submitted 2023-07-22; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitius

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neutrophil Gelatinase Associated Lipocalin and Kidney Injury Molecule-1
  Interventions: Diagnostic Test: Neutrophil Gelatinase and Kidney Injury Molecule-1

INTERVENTIONS:
Diagnostic Test: Neutrophil Gelatinase and Kidney Injury Molecule-1 — To assess Neutrophil Gelatinase associated Lipocalin and Kidney Injury Molecule-1 as biomarkers of acute kidney injury in children with Diabetic Ketoacidosis

SUMMARY:
Type 1 diabetes mellitus (T1DM) is a common, chronic, metabolic disorder that has significant consequences for physical and emotional development . The incidence of TIDM is steadily increasing in nearly all parts of the world by about 2-5% per year . Diabetic ketoacidosis (DKA) is the most serious complication of TIDM and results from metabolic abnormalities due to a severe deficiency of insulin or insulin effectiveness. Similar to diabetes, DKA has an increasing incidence and more frequently occurs in children.

DKA occurs in 20-40% of children with new-onset diabetes and in children with known diabetes who omit insulin doses or who do not successfully manage during intercurrent illness (1). Although the inpatient mortality rates of DKA are generally very low (5, 6) ,DKA is the leading with TIDM (7). DKA is associated with numerous acid-base, hydration and electrolyte derangements. Accompanied by both volume depletion and subsequent massive fluid-rehydration treatment upon presentation, children with DKA potentially have a high risk for acute kidney injury (AKI). For decades, nonconsensual definitions of AKI were used, making it difficult to obtain an accurate evaluation of the epidemiological studies

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is a common, chronic, metabolic disorder that has significant consequences for physical and emotional development. The incidence of TIDM is steadily increasing in nearly all parts of the world by about 2-5% per year. Diabetic ketoacidosis (DKA) is the most serious complication of TIDM and results from metabolic abnormalities due to a severe deficiency of insulin or insulin effectiveness. Similar to diabetes, DKA has an increasing incidence and more frequently occurs in children .

DKA occurs in 20-40% of children with new-onset diabetes and in children with known diabetes who omit insulin doses or who do not successfully manage during intercurrent illness . Although the inpatient mortality rates of DKA are generally very low ,DKA is the leading with TIDM. DKA is associated with numerous acid-base, hydration and electrolyte derangements. Accompanied by both volume depletion and subsequent massive fluid-rehydration treatment upon presentation, children with DKA potentially have a high risk for acute kidney injury (AKI). For decades, nonconsensual definitions of AKI were used, making it difficult to obtain an accurate evaluation of the epidemiological studies During the last decade, three definitions of AKI have been developed, and it is now possible to identify patients at high risk of AKI. A recent study revealed that a high proportion of children with DKA develop AKI. However, AKI remains poorly reported in children with DKA . Therefore, this study aimed to investigate the clinical characteristics and risk factors for AKI in children with DKA, and to find the risk factors of AKI on admission.

Diabetic kidney disease (DKD) is the leading cause of end-stage kidneydisease (ESKD) and dialysis in the developed world. DKD is characterizednot only by glomerular disease but also tubulointerstitial injury with tubular basement membrane thickening, tubular hypertrophy,epithelial-mesenchymal transition, glycogen accumulation andinterstitial inflammation. Although glomerular changes in diabeteshave received significant attention from researchers and clinicians,tubulointerstitial injury is known to better associate with kidney dysfunction. In fact, tubular proteinuria may precede microalbuminuriain type 1 diabetes (T1D), suggesting that tubular damage may be anearly injury pattern of DKD.4 High glucose states, such as DKA, havebeen shown to induce proximal tubular degeneration and interstitialfibrosis in both mice and humans.

More than one third of T1D youth enrolled in the SEARCH forDiabetes in Youth study had diabetic ketoacidosis (DKA) at diagnosisand in another Colorado-based study, about 55% of youth with newdiagnosis of T1D presented with DKA, which is more frequent thanwhat has been reported in international registries. Although acutekidney injury (AKI) secondary to dehydration is a well-recognizedcomplication of DKA, tubular injury attributed to DKA is poorlydescribed.5 Pathophysiologic pathways in early DKD are thought toinvolve elevated serum uric acid (SUA) and vasopressin, which are also implicated in DKA. Indeed, elevated SUA and vasopressin concentrationshave both shown to induce tubulointerstitial injury.

If DKA at diagnosis of T1D in youth is associated withtubulopathy, interventions that preserve tubular health may mitigatekidney damage. Targeted early interventions are especially importantas development of tubular injury may confer increased risk of chronickidney disease (CKD) and ESKD in the setting of DKA and AKI.

Accordingly, our study sought to assess the extent of tubular injury in DKA by characterizing the trajectories of tubular injury biomarkersover 3 months in youth with T1D diagnosed with DKA and to examinethe relationship of vasopressin and SUA in the hypothesized tubularinjury. Acute kidney injury is usually diagnosed with serialmeasurements of creatinine, cystatin C and estimated glomerular filtrationrate (eGFR) Since these parameters are influenced by iatrogenicfactors relevant to DKA care (e.g., intravenous hydration andinsulin) and are not specific for tubulointerstitial injury, we also measuredthe following tubular injury markers: neutrophil gelatinaseassociatedlipocalin (NGAL), kidney injury molecule 1 (KIM-1),chitinase 3-like 1 (YKL-40), interleukin 18 (IL-18), and monocytechemoattractant protein-1 (MCP-1).

ELIGIBILITY:
Inclusion Criteria:

* All patients with diabetic ketoacidosis below 18 years whether first time or recurrent ketoacidosis with either increase in serum creatinine more than or equal 0.3 mg/dl within 48hrs or to more than or equal 1.5 times or more baseline within 7 days or urine output less than 0.5 mL/kg/h for 6 hours.(22)

Exclusion Criteria:

* Patients with known renal disease before first attack of diabetic ketoacidosis

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - All patients with diabetic ketoacidosis below 18 years
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
biomarkers | 1 years
  To assess Neutrophil Gelatinase associated Lipocalin and Kidney Injury Molecule-1 as biomarkers of acute kidney injury in children with Diabetic Ketoacidosis

IPD SHARING:
Plan to Share IPD: No
Neutrophil Gelatinase Associated Lipocalin and Kidney Injury Molecule-1 As Biomarkers of AKI in Children With DKA

REFERENCES:
- [Background] Bjornstad P, Lanaspa MA, Ishimoto T, Kosugi T, Kume S, Jalal D, Maahs DM, Snell-Bergeon JK, Johnson RJ, Nakagawa T. Fructose and uric acid in diabetic nephropathy. Diabetologia. 2015 Sep;58(9):1993-2002. doi: 10.1007/s00125-015-3650-4. Epub 2015 Jun 7. PMID 26049401
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26049401/